CLINICAL TRIAL: NCT02685098
Title: A Clinical and Histological Analysis of Mesenchymal Stem Cells in Amputation
Acronym: CHAMP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael Murphy, MD, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1505714405
Record Dates: First submitted 2016-02-02; First posted 2016-02-18 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Ischemia; Peripheral Arterial Disease; Peripheral Vascular Disease; Vascular Disease; Arterial Occlusive Disease; Arteriosclerosis; Atherosclerosis; Cardiovascular Disease; Pathologic Processes; Orthopedic Procedures; Amputation
Keywords: Stem cells; MSCs; Mesenchymal; Amputation; BKA; below knee amputation; CHAMP; AKA; Above Knee Amputation; Stromal cells; bone marrow stem cell injection; Allogeneic
MeSH Terms: conditions — Ischemia; Peripheral Arterial Disease; Peripheral Vascular Diseases; Vascular Diseases; Arterial Occlusive Diseases; Arteriosclerosis; Atherosclerosis; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Active/Treatment Group (Experimental): Amputation performed at 7 days post allogeneic bone marrow derived mesenchymal stem cell injections.
  Interventions: Biological: Allogeneic bone marrow derived mesenchymal stem cells
- Observation Group 1 (No Intervention): Amputation performed with no MSC administration. Subjects will be followed for incidence of infection and wound healing status to week 24 as a comparator to the Active/Treatment group.
- Observation Group 2 (No Intervention): Tissue Collection Group:
  Amputation performed with no MSC administration. Subjects will not be followed after amputation is performed. Tissue collection will occur at time of amputation.
- Observation Group 3 (No Intervention): Patients undergoing lower extremity bypass grafting procedure. Skeletal muscle samples of the sartorius and anterior tibial muscle will be collected for comparison to treatment group. No study testing, nor follow up visits will occur.
- Control Group 4 (No Intervention): Patients undergoing a standard of care surgical procedure under anesthesia. Core needle biopsies will be collected from the anterior tibial muscle at the time of surgical procedure. No study testing, nor follow up visits will occur.

INTERVENTIONS:
Biological: Allogeneic bone marrow derived mesenchymal stem cells — Injection of HLA-A2+ and/or gender mismatched allogeneic MSCs above the site of amputation and into the anterior tibialis muscle (ATM) of patients scheduled for semi-elective lower extremity major amputation at 7 days before amputation.
  Other Names: cBMA; MSCs
  Arms: Active/Treatment Group

SUMMARY:
Patients undergoing semi-elective lower extremity major amputation from complications associated with atherosclerotic limb ischemia will received intra-muscular injections of allogeneic Mesenchymal Stromal Cells in the leg above and below the point of amputation to prevent ischemic wound complications after surgery and decrease the incidence of revision and further amputation. Cohort Groups 1-4 will serve as controls.

DETAILED DESCRIPTION:
This is a phase I single center open label trial study that will enroll twenty-six (26) patients requiring semi-elective lower extremity major amputation within a 30 day period for non-infectious complications related to critical limb ischemia (CLI). After enrollment patients will be scheduled for amputation 7 days after MSC administration. The investigational treatment uses allogeneic bone marrow derived mesenchymal stem cells at the point of care. Allogeneic MSCs will be injected in the gastrocnemius muscle and anterior tibialis muscle of twenty-six (26) patients undergoing major amputation. Through a review of treatment related adverse events over 6 months we will test the hypothesis that allogeneic MSCs do not result in significant cardiovascular, respiratory, or infectious treatment related adverse events. Through an exploratory investigation we will assess the efficacy of MSCs in promoting freedom from gangrene, revision of amputation, and death after major amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 40 and ≤90 years of age.
2. Patients requiring lower extremity major amputation, as determined by an independent vascular specialist.
3. If ulceration or gangrene present, it is distal to malleoli (to allow adequate length of ATM area of approximately 3cm x 10cm x 3 cm)
4. Amputation can safely be performed up to 30 days after screening, as determined by an independent vascular or orthopedic surgeon.
5. Females of childbearing potential must be willing to use one form of birth control for the duration of the study. Female participants must undergo a blood or urine pregnancy test at screening.

Exclusion Criteria:

1. Patients who are pregnant, planning to become pregnant in the next 12 months, or lactating.
2. CHF hospitalization within the last 1 month prior to enrollment.*
3. Acute coronary syndrome in the last 1 month prior to enrollment.*
4. HIV positive, or active, untreated HCV as determined by review of medical records.
5. History of cancer within the last 5 years, except basal cell skin carcinoma
6. Inability to provide written informed consent due to cognitive or language barriers (interpreter permitted).
7. Concurrent enrollment in another clinical investigative trial that may alter the outcomes of enrollment in this trial.
8. Any condition requiring immunosuppressant medications (e.g., for treatment of organ transplants, psoriasis, Crohn's disease, alopecia areata).
9. Presence of any clinical condition that in the opinion of the PI or the sponsor makes the patient not suitable to participate in the trial.

   * As defined by the standard definitions of CHF and ACS by the American Heart Association.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events occurring during the enrollment period as assessed by the Investigator using the MeDRA scale. | Primary follow up in a 6 month period
  Treatment-related adverse events will be categorized in overlapping systems of cardiovascular, respiratory, or infectious and severities of serious adverse events (SAE) and major adverse cardiac events (MACE). The sum and difference between routes of delivery will be reported. Confidence intervals will be generated and summarize the data by the method of the Wilson Score Interval. Binomial confidence intervals at the 95% confidence level and p-values for these groups will be calculated. Continuous confidence intervals at the 95% level will be constructed to explore the effect of administration of MSCs on the composite endpoint at 6-months of death, amputation revision and gangrene, and will be compared to historical cohorts. The critical levels for the multiplicity adjustment will be determined by simple Monte Carlo simulation.Unanticipated SAEs and those affecting the rights, safety, or welfare of subjects will be documented and reported immediately upon discovery.

SECONDARY OUTCOMES:
Gene and protein arrays, IHC staining, and multiparametric flow cytometry will measure the time period of retention of allogeneic MSCs in harvested human skeletal muscle tissue post-MSC implantation. | Primary follow up in a 6 month period
  Quantities over time of MSC will be fit to an exponential decay curve using a residual pseudo-likelihood procedure and cell half-life (λ) will be estimated. Binomial confidence intervals at the 95% confidence level and p-values will be calculated for the presence or absence of MHC expression and SDF-1activation. The correlation between capillary density (CD31 counts) with tissue perfusion (ICA) for each time point will be estimated by Spearman's rank coefficient. The gene and protein expression profiles and histological findings will be used to test the hypotheses that MSCs have limited survival post-injection.
Recruitment of proangiogenic hematopoietic cells into sites of ischemia will be measured and reported as assessed by the role of MSCs injected in human skeletal muscle at the time of amputation. | Primary follow up in a 6 month period
  Continuous confidence intervals at the 95% level will be constructed to explore differences among the time-tiered administration of MSC for (1) the CD34+CD133+ pro-angiogenic hematopoietic cells recruitment of HIF-1α/SDF-1/CXCR4 to ischemic muscle, (2) the quantify of capillary density in muscle fibers using hematoxylin phloxin saffron and CD31 counts, (3) VEGF-A,C,D, hepatocyte growth factor, angiopoietin-1 to characterize angiogenic cytokine expression, (4) percent coverage, fiber diameter and cross-sectional area to examine changes in morphology. The gene and protein expression profiles and histological findings will be used to test the hypotheses that MSCs act to recruit CD34+CD133+ proangiogenic hematopoietic cells.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Murphy, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy MP, Lawson JH, Rapp BM, Dalsing MC, Klein J, Wilson MG, Hutchins GD, March KL. Autologous bone marrow mononuclear cell therapy is safe and promotes amputation-free survival in patients with critical limb ischemia. J Vasc Surg. 2011 Jun;53(6):1565-74.e1. doi: 10.1016/j.jvs.2011.01.074. Epub 2011 Apr 22. PMID 21514773
- [Derived] Wang SK, Green LA, Drucker NA, Motaganahalli RL, Fajardo A, Murphy MP. Rationale and design of the Clinical and Histologic Analysis of Mesenchymal Stromal Cells in AmPutations (CHAMP) trial investigating the therapeutic mechanism of mesenchymal stromal cells in the treatment of critical limb ischemia. J Vasc Surg. 2018 Jul;68(1):176-181.e1. doi: 10.1016/j.jvs.2017.09.057. Epub 2018 Feb 1. PMID 29395424